CLINICAL TRIAL: NCT02917291
Title: Clinical Trial of Phase 1/2 to Evaluate the Feasibility, Safety, Tolerability and Preliminary Efficacy of the Administration of FAB117-HC, a Drug Whose Active Ingredient is HC016, Allogeneic Adipose Derived Adult Mesenchymal Stem Cells Expanded and Pulsed With H2O2, in Acute Traumatic SCI Patients.
Brief Title: Safety and Preliminary Efficacy of FAB117-HC in Patients With Acute Traumatic Spinal Cord Injury
Acronym: SPINE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ferrer Internacional S.A. (Industry)
Collaborators: Histocell, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAB117-CT-01
Record Dates: First submitted 2016-09-20; First posted 2016-09-28 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Acute Traumatic Spinal Cord Injury
Keywords: Trauma Spinal Cord; Thoracic Acute Spinal Cord Injury; Neurosurgery; Cell Therapy; ATMP; HC016 adipose mesenchymal stem cell; SPINE
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FAB117-HC (Ph 1) (Experimental): Patients with acute traumatic spinal cord injury grading AIS A (8 patients)
  Interventions: Drug: FAB117-HC
- Control group (Ph 2) (Other): Patients with acute traumatic spinal cord injury grading AIS A or B (up to 20 patients)
  Interventions: Other: Control group
- FAB117-HC (Ph 2) (Experimental): Patients with acute traumatic spinal cord injury grading AIS A or B (up to 20 patients)
  Interventions: Drug: FAB117-HC

INTERVENTIONS:
Drug: FAB117-HC — (Ph 1) Intramedullary administration. Open label dose escalation, 3 patients in cohort 1 (20 million cells) and 5 patients in cohort 2 (40 million cells)
  Arms: FAB117-HC (Ph 1)
Other: Control group — (Ph 2) No treatment will be administered
  Arms: Control group (Ph 2)
Drug: FAB117-HC — (Ph 2) Intramedullary administration of the maximum tolerated dose (20 or 40 million cells)
  Arms: FAB117-HC (Ph 2)

SUMMARY:
The main objective of the study is the evaluation of the safety and tolerability of FAB117-HC (a medicinal product containing human allogeneic adipose derived adult mesenchymal stem cells expanded and pulsed with H2O2, HC016 cells) administered at a single-time point to patients with acute thoracic traumatic spinal cord injury (SCI). The study will also include initial exploration of potential clinical efficacy. Dose levels of 20 million and 40 million cells will be administered.

DETAILED DESCRIPTION:
FAB117-HC is an investigational medicinal product whose active substance is HC016, allogeneic adipose-derived adult mesenchymal stem cells expanded and pulsed with H2O2.

The main purpose of this study is to evaluate the safety and tolerability of a single administration of FAB117-HC using: a) two sequential escalating doses administered between 72 and 120 hours post-injury, to patients with acute traumatic SCI with ASIA Impairment Scale (AIS) grade A; and b) the determined maximum tolerated dose administered up to 96 h post-injury to patients with AIS grading of A or B. The study includes also initial exploration of efficacy.

Treatment is administered by intramedullary injection into the injured spinal cord, during the decompression and stabilization surgery (DSS) of the fracture. DSS is routinely performed on almost all SCI patients.

The study has been divided into two phases:

Phase 1 (open label): 8 AIS A patients with lesion located between D1 and D12 will be included in 2 sequential cohorts.

Phase 2 (randomized, controlled, double-blind): Up to 40 AIS A or B patients with lesion located between D1 and D12, will be randomly divided into two groups (control and treated) that will be balanced in AIS grade.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 (2 Cohorts)

1. Male or female subjects ≥ 16 to ≤ 70 years.
2. ASIA impairment grade A.
3. Either a level of injury between D1-D12 both inclusive (cohorts 1 and 2).
4. Single traumatic spinal cord injury as defined by MRI.
5. Injury occurred between 72 and 120h before undergoing DSS and treatment.
6. Clinically and haemodynamically stable, under medical criteria, enough to undergo DSS.
7. Able to give informed consent either in writing or orally in the presence of a witness.

Phase 2 (2 Groups)

1. Male or female subjects ≥ 16 to ≤ 70 years.
2. ASIA impairment grade A or B.
3. An injury between D1 and D12, both inclusive.
4. Single traumatic spinal cord injury as defined by MRI.
5. Injury occurring up to 96 h before undergoing DSS and treatment.
6. Clinically and haemodynamically stable enough, under medical criteria, to undergo DSS.
7. Able to give informed consent either in writing or orally in the presence of a witness.

Exclusion Criteria:

1. Participated in a previous clinical study and received an investigational product within 28 days of SCI (within 5 years of SCI if the investigational product is a cell-based medicine).
2. Radiological or MRI or DSS evidence of complete or partial spinal cord transection.
3. Inability to unequivocally identify the injection sites.
4. Multiple injuries to the neurological spinal cord at different levels.
5. Patients with any of these additional conditions:

   1. Penetrating spinal cord injuries.
   2. Associated trauma or injury to the brachial and / or lumbosacral plexus.
6. Active infection in the surgical area.
7. Haemodynamic instability contraindicating DSS procedure in the time frame defined for inclusion in the trial.
8. Multiple organ failure.
9. Severe multiple trauma that hampers the stabilization procedure in the defined term for the inclusion in the trial.
10. Significant head injury (Score on the Glasgow scale less than or equal to 13 and / or abnormal MRI/CT, meaning oedema, axonal lesion and/or haemorrhage) or other injury that in the investigator's opinion is sufficient to interfere with the assessment of spinal cord function or compromise the validity of patient data.
11. Patients undergoing mechanical ventilation that does not allow a prior clinical examination.
12. Inability to communicate with the neurological examiner so that the validity of patient data could be unreliable.
13. Coma or significant impairment in the level of consciousness, including unconsciousness due to sedative-analgesic medications, that interferes with the performance or interpretation of assessments specific in the protocol.
14. Preexisting or current significant diseases such as hepatitis C, HIV, epilepsy, neoplastic disease or other diseases that could cause neurological deficits including syphilis, myelopathy, and polyneuropathy.
15. Background or acute episode of Guillain-Barre syndrome.
16. History of meningitis or meningoencephalitis.
17. Current autoimmune disease treated with immunosuppressant therapy.
18. Patients with history of severe thrombophilia or under anticoagulant pharmacological therapy which long elimination half-live prevents a rapid transition to heparin (like dabigatran and rivaroxaban).
19. Presence of any psychiatric illness, as defined by the DSM-IV-TR, or medically unstable illness that means a hindrance to the adherence to rehabilitation and/or to the informed consent signature.
20. Pregnant women or women of childbearing age who are not using an appropriate method of contraception and, moreover, are not willing to continue to use it for the duration of the trial. If the patient is menopausal or sterile, it must be documented in the medical record.
21. Women who are breastfeeding if unwilling to stop at the time of recruitment.
22. History of allergy with anaphylactic shock.
23. Patients with known hypersensitivity to any of the excipients of FAB117-HC.
24. Patients with known hypersensitivity to penicillin, streptomycin, enzymes (trypsin or collagenase), bovine serum or DMSO.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability of a single dose of FAB117-HC when administered by intramedullary injection into the injured spinal cord | One year

SECONDARY OUTCOMES:
Changes in neurological function using the International Standards for Neurological Classification of SCI (ISNCSCI) scale, examinations at 24h, 72h, 7d, 14d, 28d, 90d and 360 days after injection of FAB117-HC | One year
Changes in the functional assessment of Spinal Cord Independence Measure (SCIM III) | Day 28 and Day 90
Changes in Somatosensory-Evoked Potentials (SSEP) electrophysiological assessment test. | Day 28 and Day 90
Changes in Motor-Evoked Potentials (MEP) electrophysiological assessment test | Day 28 and Day 90

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Complejo Hospitalario de Toledo (HNP y VS), Toledo
  - Hospital Universitari La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza